CLINICAL TRIAL: NCT06663839
Title: A Phase I, Open-label, Dose Finding Study of NILK-2301, a Bispecific CEACAM5 X CD3 Engaging Antibody, in Patients with Locally Advanced or Metastatic Low Tumor Volume (LTV) Colorectal Cancer
Brief Title: A Study of NILK-2301 in Patients with Locally Advanced or Metastatic Low Tumor Volume (LTV) Colorectal Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Light Chain Bioscience - Novimmune SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCB-2301-001; 2023-508058-24-01 (EU CTIS Number)
Record Dates: First submitted 2024-10-25; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer Metastatic
Keywords: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NILK-2301 Single Agent (Experimental): NILK-2301 will be evaluated in patients with locally advanced or metastatic low tumor volume colorectal cancer
  Interventions: Drug: Biological NILK-2301

INTERVENTIONS:
Drug: Biological NILK-2301 — Treatments will be administered every two weeks in 28-day cycles for up to 12 months until disease progression, unacceptable toxicity, or Investigator/patient decision to withdraw study consent. Should evidence emerge showing that treatment beyond one year may prolong benefit in responding patients, the protocol will be amended to ensure that these responding patients may continue with the study treatment beyond 12 months until disease progression.

SUMMARY:
Study LCB-2301-001 is an open-label, Phase 1, dose escalation (Part A) and expansion (Part B), first-in-human clinical study of NILK-2301 in patients with locally advanced or metastatic low tumor volume (LTV) colorectal cancer.

The dose escalation part (Part A) of the study will evaluate the safety and tolerability of escalating doses of NILK-2301 to determine the maximum tolerated dose (MTD) and non-tolerated toxic dose (NTD) of NILK-2301 monotherapy. The expansion part (Part B) will further evaluate the safety and efficacy of NILK-2301 monotherapy administered at or below the MTD in up to 10 additional subjects in order to determine the recommended Phase 2 dose (RP2D).

Treatments will be administered every two weeks in 28-day cycles for up to 12 months until disease progression, unacceptable toxicity, or Investigator/patient decision to withdraw study consent.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ≥ 18 years of age at the time of signing the informed consent form (ICF).
2. Histologically or cytologically confirmed diagnosis of CRC.
3. Patients with locally advanced or metastatic disease

   * after at least 1 prior systemic treatment for the primary malignancy
   * and who have failed treatment with, are intolerant to, or are not candidates for available therapies that are known to confer a clinical benefit to patients with these tumor entities.
4. Measurable disease according to the revised RECIST guideline version 1.1 (5).
5. Tumor lesions of up to approximately 50 cc estimated with the sum of all measurable lesions (excluding pathological lymph nodes) longest diameter (SLD). SLD should be < 7 cm.
6. Any measurable lesion (excluding pathological lymph nodes) longest diameter ˂ 5 cm.
7. Eastern Cooperative Oncology Group performance status (ECOG PS) 0-1.
8. Subjects must have the following laboratory values (determined by local lab):

   * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L, the use of colony- stimulating factors, i.e., granulocyte colony-stimulating factor (G-CSF) or GM-CSF, within 14 days before the test is not allowed.
   * Platelets ≥ 100 x 109/L, transfusion support within 14 days before the test is not allowed.
   * Hemoglobin ≥ 10 g/dL. Prior RBC transfusion is permitted.
   * Potassium within normal limits or correctable with supplements.
   * Aspartate aminotransferase (AST), alanine aminotransferase (ALT) ≤ 2.5 x upper limit of normal (ULN), or Alkaline Phosphatase (ALP) ≤ 3 × ULN
   * Serum bilirubin < 1.5 x ULN.
   * Calculated glomerular filtration rate of ≥ 45 mL/min/1.73 m2, according to the MDRD abbreviated formula.
   * International normalized ratio (INR) < 1.5 x ULN and partial thromboplastin time (PTT)< 1.5 x ULN.
9. Females of childbearing potential (FCBP) must:

   * have two negative urine or serum pregnancy tests as verified by the Investigator prior to starting NILK-2301; the subject may not receive NILK-2301 until the Investigator has verified that the result of the pregnancy test is negative. A urine or serum pregnancy test is required at screening and within 72 hours prior to dosing on Cycle 1, Day 1, and within 72 hours prior to Day 1 of every subsequent cycle. Note: the Cycle 1, Day 1 pregnancy test does not need to be repeated if the screening pregnancy test was done within 72 hours prior to dosing. A serum or urine pregnancy test (Investigator's discretion) must also be performed at the end of study for each FCBP; and
   * agree to use and be able to comply with a highly effective birth control method, i.e., one that can achieve a failure rate of less than 1% per year when used consistently and correctly, from signing the ICF, throughout the study, and for up to 28 days following the last dose of NILK-2301

Exclusion Criteria:

1. Patient has known hypersensitivity to NILK-2301 or any of the constituent compounds.
2. Patients with CNS lesions and / or bone disease.
3. Patients with pleural and / or pericardial tumor lesions.
4. Radiotherapy to the target lesions within 4 weeks prior to the first NILK- 2301 infusion.
5. Prior anti-cancer therapy including chemotherapy, hormonal therapy, and investigational agents within 28 days prior to starting NILK-2301 dosing. Note: low dose steroids (oral prednisone or equivalent ≤ 10 mg per day, including systemic or topic use), localized non-central nervous system (CNS) radiotherapy of non-target lesions, and treatment with bisphosphonates and RANKL inhibitors are not criteria for exclusion.
6. Other investigational therapies must not be used, i.e., treatment within another clinical trial is not permitted, while the patient is on study. COVID- 19 vaccination is allowed only starting from Cycle 2 (if not completed before study inclusion).
7. Severe cardiac dysfunction (NYHA classification III-IV).
8. Significant hepatic dysfunction (serum bilirubin ≥ 1.8 mg/dL or AST and/or ALT ≥ 2.5 times ULN), or ALP ≤ 3 × ULN.
9. Patients with known human immunodeficiency virus (HIV) infection or known history or serological evidence of hepatitis B or C virus infection.
10. Uncontrolled active systemic bacterial, viral, fungal, or other infection (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment), or intravenous anti-infective treatment within 2 weeks prior to first dose of NILK-2301.
11. Confirmed history or current autoimmune disease or other diseases or conditions resulting in permanent immunosuppression or requiring permanent immunosuppressive therapy. Low- dose steroids (oral prednisone or equivalent ≤ 10 mg per day) for rheumatoid arthritis or similar conditions are allowed.
12. Patients with concomitant active malignancy requiring ongoing systemic treatment.
13. Patients with CNS metastases, history of leptomeningeal disease, or seizure disorder requiring therapy (e.g., steroids or anti-epileptics).
14. ANC < 1 x 109/L (the use of colony stimulating factors, G-CSF or GM-CSF, within 14 days before the test is not allowed).
15. Pregnancy and lactation.
16. History of psychiatric illness or substance abuse likely to interfere with ability to comply with protocol requirements or give informed consent.
17. Significant medical diseases or conditions, including laboratory abnormalities, as assessed by the Investigators and Sponsor, that would substantially increase the risk-benefit ratio of participating in the study. This includes, but is not limited to, myocardial infarction within the last 6 months, unstable angina or unstable life-threatening arrhythmias, uncontrolled diabetes mellitus, severely immunocompromised state, and major surgery ≤ 4 weeks prior to starting NILK-2301.
18. Patients in whom acute toxic effects of any prior radiotherapy, chemotherapy, or surgical procedure have not resolved to Grade ≤ 1 or returned to baseline except for alopecia (any grade), anemia, and peripheral neuropathy (for the latter, recovery to Grade ≤ 2 is acceptable).
19. Exposure to live or live attenuated vaccine within 28 days prior to signing the ICF.
20. Previous treatment with a CEACAM5 targeting agent.
21. Prior treatment with a T-cell bispecific antibody or CAR T-cells.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-04-12 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | Up to 12 months
  Is defined as any of the toxicities occurring within the DLT window (Cycle 1, Days 1 to 28) except those that are clearly and incontrovertibly due to extraneous causes.
Non-Tolerated Dose (NTD) | Up to 12 months
  Is defined as a dose level at which 2 or more of up to 6 evaluable patients in a cohort experience a DLT in the 4-week DLT window.
Maximum Tolerated Dose (MTD) | Up to 12 months
  Is defined as the last cohort below the NTD with 0 or 1 out of 6 evaluable subjects experiencing a DLT during the 4-week DLT window.
Adverse Events (AEs) | Up to 12 months
  Number of patients with AEs as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | Up to 12 months
  Is defined as the time from the first dose of NILK-2301 to progressive disease or death from any cause, whichever occurs first
Overall Survival (OS) | Up to 12 months
  Is defined as the time from the first dose of NILK-2301 to death from any cause
Pharmacokinetics - Cmax | Up to 12 months
  Maximum concentration of drug
Presence of anti-drug antibodies (ADA) | Up to 12 months
  Detection of ADAs in patients

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - START Madrid-FJD, Hospital Fundación Jiménez Díaz, Madrid

IPD SHARING:
Plan to Share IPD: No